CLINICAL TRIAL: NCT03242720
Title: Effects of Positive Airway Pressure on Atrial Fibrillation Recurrence Risk After Catheter Ablation in Patients With Atrial Fibrillation and Obstructive Sleep Apnea-A Pilot Randomized Controlled Trial
Brief Title: Effects of PAP on Afib Recurrence Risk After Catheter Ablation in OSA Patients
Acronym: OSA-AFIB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Clete A. Kushida, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 41798
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Obstructive Sleep Apnea; Atrial Fibrillation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Positive Airway Pressure (Active Comparator): Active positive airway pressure for treatment of Obstructive Sleep Apnea
  Interventions: Procedure: Cardiac Ablation for Atrial Fibrillation
- Sham Positive Airway Pressure (Sham Comparator): Sham positive airway pressure for treatment of Obstructive Sleep Apnea
  Interventions: Procedure: Cardiac Ablation for Atrial Fibrillation

INTERVENTIONS:
Procedure: Cardiac Ablation for Atrial Fibrillation — Ablation of arrhythmia focus in the heart for atrial fibrillation

SUMMARY:
With this pilot study, we are hoping to test the feasibility of a larger study in the future and to learn whether positive airway pressure therapy reduces the recurrence risk of atrial fibrillation after successful catheter ablation procedure among patients with atrial fibrillation and obstructive sleep apnea. The results from this study will help us refine the design for a future larger study, and will ultimately improve care of patients with obstructive sleep apnea and atrial fibrillation.

DETAILED DESCRIPTION:
Obstructive sleep apnea, a sleep-related breathing disorder in which breathing stops for short periods during sleep, is a common condition in patients with atrial fibrillation. Studies have shown that up to 75% of atrial fibrillation patients undergoing catheter ablation procedure have obstructive sleep apnea. Obstructive sleep apnea increases the risk of atrial fibrillation recurrence after successful catheter ablation by 40%. However, whether treatment of obstructive sleep apnea with positive airway pressure (PAP, the current most effective treatment for obstructive sleep apnea that uses a machine to help breathe more easily) reduces the risk of atrial fibrillation recurrence is not fully understood. The purpose of this study, therefore, is to examine whether positive airway pressure therapy reduces atrial fibrillation recurrence after catheter ablation in patients with obstructive sleep apnea and atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years or older
2. First-time catheter ablation for atrial fibrillation
3. Moderate-to-severe obstructive sleep apnea diagnosed with a sleep study (apnea-hypopnea index ≥ 15)

Exclusion Criteria:

1. Current or prior use of positive airway pressure for obstructive sleep apnea
2. Any household member with current/past positive airway pressure use
3. Did not meet minimal adherence to positive airway pressure treatment (≥ 4 hours/night and ≥ 70% of time in 2 weeks)
4. History of motor vehicle or occupational accident related to excessive sleepiness
5. Severe nocturnal desaturation documented on sleep study as >10% of total sleep time with oxygen saturation of < 75%
6. Any condition determined by physicians that constrains the use of positive airway pressure such as anatomically fixed nasal obstruction, neurological impairment, and significant claustrophobia.
7. Congestive heart failure (New York Heart Association IV)
8. Severe valvular disease
9. Planned coronary revascularization procedure in the next 6 months
10. Severe pulmonary disease
11. Participation in another treatment intervention trial that might influence results of this trial
12. Ablation procedure scheduled in the next 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation recurrence | 6 months after ablation
  Risk of Atrial Fibrillation recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Clete A Kushida, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Sleep Medicine Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No